CLINICAL TRIAL: NCT01625741
Title: Phase II Study of High-Dose Rituximab in High-Risk Chronic Lymphocytic Leukemia Patients in Suboptimal Response After Induction Immunochemotherapy
Acronym: HYDRIC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Stopped by Principal Investigator decision
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HYDRIC
Record Dates: First submitted 2012-06-06; First posted 2012-06-21 (Estimated); Last update posted 2015-09-29 (Estimated); Status verified 2015-09

CONDITIONS: Chronic Lymphocytic Leukemia
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- rituximab (Experimental): 4 monthly administrations of rituximab
  Interventions: Drug: Rituximab

INTERVENTIONS:
Drug: Rituximab — 2000 mg, IV, monthly, for 4 months (= 4 doses)
  Other Names: Mabthera

SUMMARY:
This study explores the potential to improve the quality of response obtained after induction treatment in Chronic Lymphocytic Leukemia (CLL), by giving a short and intense consolidation schema using high-dose rituximab. Patients in suboptimal response (Minimal Residual Disease persistence) after induction will be selected, as well as those who have a Minimal Residual Disease (MRD) relapse after having achieved MRD negativity.

DETAILED DESCRIPTION:
This study is reserved for patients with residual disease at the end of therapy at the level of Minimal Residual Disease (MRD-positive either in the peripheral blood at least 6 months after the last dose of rituximab-containing immunochemotherapy or in the bone marrow at least 3 months after the last dose of rituximab-containing immunochemotherapy). Patients who have achieved MRD eradication and who have MRD relapse (reappearance of residual leukemic cells using 7/8-color flow cytometry in peripheral blood or bone marrow) are also eligible for the study.

Rituximab will be given intravenously at a monthly dose of 2000 mg four months (in total 4 doses of 2000 mg each), starting within one month after informed consent signature.

The patients will be followed during the treatment period with rituximab. A final evaluation will be done 3 months after the last dose of rituximab.

ELIGIBILITY:
Inclusion Criteria:

* B-cell Chronic Lymphocytic Leukemia defined by standard NCI criteria in first line or in relapse
* > 18 years-old
* Presence of Minimal Residual Disease (MRD positivity) by Flow Cytometry criteria in these two clinical situations :

  1. Patients in Complete Remission (defined by standard criteria including Bone Marrow examination) after rituximab-containing immunochemotherapy (ICT), who show persisting MRD either in the Peripheral Blood at least 6 months after the last dose of rituximab-containing immunochemotherapy or in the Bone Marrow at least 3 months after the last dose of rituximab-containing ICT
  2. Patients in continuous CR who show MRD relapse in PB or BM without clinical progression (as defined by NCI) at any time after ICT
* ICT should have comprised:

  1. Rituximab combined with fludarabine, with or without an alkylating drug, with or without an anthracycline (ex: Fludarabine-Rituximab, Fluda-Cyclophsphamide-Rituximab, FCR-Mitoxantrone, R-bendamustine…)
  2. At least 4 cycles
* Patients should have recovered from the toxicities of ICT
* POOR PROGNOSTIC FEATURES (before induction ICT) defined by at least one of the following markers: stage C Binet, unmutated IgVH genes, 17p deletion, 11q deletion, Zap-70 positivity, high CD38, mutated IgVH genes if VH3-21 usage
* In addition, in patients with 11q deletion and/or presence of bulky lymph nodes prior to induction therapy, absence of profound lymph nodes at response evaluation should have been confirmed by CT scan
* CIRS ≤6
* Absence of significant geriatric syndromes and/or significant limitations in instrumental activities of daily living (IADL)
* Performance status (ECOG) < 2
* Neutrophils > 1000/microL, platelets > 100,000/microL
* Creatinine clearance > 50 ml/min (clearance can be reevaluated after adequate hydration of the patient)
* Patient's written informed consent

Exclusion Criteria:

* Less than CR defined by standard criteria response after ICT
* Ongoing active infections (bacterial, viral or fungal)
* Known infection with HIV
* Subjects with any serological evidence of current or past hepatitis B or hepatitis C exposure are excluded unless the serological findings are clearly due to vaccination.
* Concomitant treatment with steroids, or any immunosuppressive drug
* Uncontrolled autoimmune hemolytic anemia or thrombocytopenia
* Transformation into an aggressive B-cell malignancy (eg. diffuse large B-cell lymphoma, Hodgkin lymphoma)
* Pregnancy, breast feeding, female patients with childbearing potential or male patients who are unwilling to use adequate contraception
* Intolerance to rituximab
* Concomitant severe disease (uncompensated cardiac insufficiency, severe respiratory insufficiency…)
* Severe hypogammaglobulinemia with recurrent infections, unless the patient is receiving substitutive IV immunoglobulins
* Transaminases (AST, ALT) > 3 xULN
* Conjugated bilirubin > 2 xULN
* Prior autologous stem cell transplantation less than 12 months
* Prior allogeneic stem cell transplantation
* Central Nervous System involvement
* Any coexisting medical or psychological condition that would preclude participation to the required study procedures
* Prior history of malignancies, other than CLL, unless subject has been free of the disease for > 4 years. Exceptions include the following: basal cell carcinoma of the skin, squamous cell carcinoma of the skin, carcinoma in situ of the cervix, carcinoma in situ of the breast, incidental histologic finding prostate cancer (TNM stage of T1a or T1b)
* Participation in any clinical study or having taken any investigational therapy which would interfere with the study drug for a disease other than CLL, within 28 days prior to initiating the maintenance therapy.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2012-07; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
rate of conversion into Minimal Residual Disease negativity | Month 7 (= 3 months after the last dose of rituximab)
  Evaluate the rate of conversion into MRD negativity 3 months after the administration of 4 monthly courses of high-dose (2000 mg) rituximab in high-risk CLL patients with suboptimal response after immunochemotherapy (ICT), or MRD relapse after ICT.

SECONDARY OUTCOMES:
toxicity of the consolidation treatment by rituximab | from first administration of rituximab until end of follow-up period (= 12 months after the last rituximab administration)
Pharmacokinetic/Pharmacodynamic correlation | month 7
  correlation between the level of MRD conversion at month 7 and pharmacokinetic dosage of rituximab performed after each rituximab perfusions, 1 month and 3 months after last rituximab.
quality of life study | during 17 months
  from selection visit until last follow-up visit planned 1 years after the last rituximab perfusion

CONTACTS AND LOCATIONS:
Overall Officials: Eric Van Den Neste, MD, PhD, Principal Investigator — Cliniques universitaires Saint-Luc- Université Catholique de Louvain
Locations (15):
- Belgium (15):
  - ZNA Middelheim, Antwerp
  - Clinique Sud Luxembourg, Arlon
  - AZ Sint-Jan, Bruges
  - Clinique Saint Jean, Brussels
  - ULB Erasme, Brussels
  - Cliniques universitaires Saint Luc, Brussels
  - Grand Hôpital de Charleroi, Charleroi
  - UZ Gent, Ghent
  - Hôpital de Jolimont, Haine-Saint-Paul
  - KUL Gasthuisberg, Leuven
  - CHU ULg Sart Tilman, Liège
  - CHR Clinique Saint Joseph, Mons
  - Clinique Saint Pierre, Ottignies
  - Heilig-Hartziekenhuis, Roeselaere
  - Clinique universitaire de Mont Godinne, Yvoir